CLINICAL TRIAL: NCT05347719
Title: Virtual Mindfulness Training for Adults With History of Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clemson University (Other)
Collaborators: Prisma Health-Upstate (Other)
Responsible Party: Principal Investigator, Heidi Zinzow, Professor, Clemson University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00092709
Record Dates: First submitted 2022-04-14; First posted 2022-04-26 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Major Depressive Disorder
Keywords: Mindfulness Based Cognitive Therapy; Major Depressive Disorder; Virtual Delivery; Community Health
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: To achieve our study aims, we designed a randomized, controlled trial with a treatment as usual (TAU) control group. A total of 240 eligible participants will be randomized to either an MBCT intervention group (Group 1) or an TAU control (Group 2). In Phase I, Group 1 will complete the intervention and Group 2 will remain in TAU. In Phase II , Group 2 will complete the intervention and Group 1 will continue TAU. Depending on the recruitment site, TAU may consist of receiving psychotherapy, pharmacotherapy, or combined treatment within an academic medical center. Data collection will be completed at baseline, post-intervention for Group 1 and pre-intervention for Group 2, and after follow-up for Group 1 and post-intervention for Group 2. This design allows us to provide fair treatment for both trial arms as well as allowing for follow-up assessment of Group 1.
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBCT Intervention (Experimental): Eight weekly two-hour mindful MBCT intervention sessions led by a trained healthcare provider. Post-intervention, the experimental group will receive treatment as usual.
  Interventions: Behavioral: MBCT Intervention
- Wait List Control (No Intervention): Participants will engage in treatment as usual during the baseline period. After the experimental group completes the MBCT intervention, the wait list control group will complete the MBCT intervention.

INTERVENTIONS:
Behavioral: MBCT Intervention — Eight weekly two-hour mindful MBCT intervention sessions involving training in mindfulness meditation and cognitive-behavioral methods. Sessions will be designed to increase participant awareness of internal reactions that trigger relapse in MDD and to provide participants with techniques to detach from dysfunctional cognitive processes and redirect their attention to experiences. Outside of the sessions, participants will be assigned daily homework exercises and provided with handouts and audio recordings of mindfulness exercises to use in their practice.
  Arms: MBCT Intervention

SUMMARY:
Mindfulness Based Cognitive Therapy (MBCT) has shown to be an effective method of preventing relapse of an episode Major Depressive Disorder (MDD). MBCT is a group program that integrates mindfulness skills training with cognitive-behavioral strategies. However, the cost of MBCT is not affordable to many families. The aim of this study is to explore the feasibility and efficacy of an MBCT intervention designed to be delivered at low cost through a virtual delivery format. This study will recruit 240 participants who are in remission from depression and randomize them to an MBCT intervention group or treatment as usual (TAU) for the wait list control group. The wait list control group will complete the intervention after the MBCT intervention group. Assessment administered at pre-intervention (baseline), post-intervention for experimental group, and post-intervention for the wait list control group and follow-up for experimental group. The primary outcome is to test the efficacy of this community-based delivery in reducing depression severity and psychiatric distress in the relapse of an episode of MDD. The secondary outcomes include perceived stress, post-traumatic stress symptoms, adherence to treatment plans not given as part of this study, frequency of relapse of MDD, mindfulness skills, and quality of life. This study will also examine the following potential moderators and correlates of intervention outcomes: comorbid diagnoses, life events history, and MBCT intervention adherence. Finally, the study will examine the following mediators of intervention outcome: mindfulness skills, emotion regulation skills, executive functioning skills, savoring, and positive and negative affect.

DETAILED DESCRIPTION:
Mindfulness Based Cognitive Therapy (MBCT) has shown to be an effective method of preventing relapse of an episode Major Depressive Disorder (MDD). MBCT is a group program that integrates mindfulness skills training with cognitive-behavioral strategies. However, the cost of MBCT is not affordable to many families. The aim of this study is to explore the feasibility and efficacy of an MBCT intervention designed to be delivered at low cost through a virtual delivery format. The study will recruit 240 participants who are in remission from depression and randomize them to an MBCT intervention group or treatment as usual (TAU) for the wait list control group. The wait list control group will complete the intervention after the MBCT intervention group. Assessments will be administered at pre-intervention (baseline), post-intervention for experimental group (week 8), and post-intervention for the wait list control group and follow-up for experimental group (week 16). The primary outcome is to test the efficacy of this community-based delivery in reducing depression severity and psychiatric distress in the relapse of an episode of MDD. The secondary outcomes include perceived stress, post-traumatic stress symptoms, adherence to treatment plans not given as part of this study, frequency of relapse of MDD, mindfulness skills, and quality of life. This study will also examine the following potential moderators and correlates of intervention outcomes: comorbid diagnoses, life events history, and MBCT intervention adherence. Finally, this study will examine the following mediators of intervention outcome: mindfulness skills, emotion regulation skills, executive functioning skills, savoring, and positive and negative affect.

ELIGIBILITY:
Inclusion Criteria:

* be over 18 years of age
* be a resident of upstate South Carolina or Prisma Health beneficiary
* have a SCID confirmed diagnosis of a prior MDD episode
* be willing to share contact information
* have English literacy 6th grade or above
* be able to attend intervention sessions.

Exclusion Criteria:

* current psychosis, dementia, moderate to severe traumatic brain injury, or active suicidality
* persistent antisocial behavior
* persistent self-injury requiring clinical management
* an acute episode of a substance use disorder episode (met two or more SUD criteria in the past two weeks, excluding for tobacco or marijuana use)
* an acute episode of MDD (met two or more MDD criteria in the past two weeks)
* an active diagnosis of Bipolar Disorder
* previously completed or currently attending a standard MBCT intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Depression Severity | Baseline, 8 weeks (post-intervention for experimental group), 16 weeks (follow-up for experimental group, post-intervention for control group)
  Depression severity will be assessed with the Patient Health Questionnaire (PHQ-9; Kroenke, Spitzer & Williams 2001). PHQ-9 scores of 5, 10, 15, and 20 represents mild, moderate, moderately severe, and severe depression.
Change in Psychiatric Distress | Baseline, 8 weeks (post-intervention for experimental group), 16 weeks (follow-up for experimental group, post-intervention for control group)
  Psychiatric distress will be measured using the depression and anxiety subscales of the Brief Symptom Inventory (BSI; Derogatis & Melisaratos,1983). Items, such as "your feelings being easily hurt," are ranked on a 5-point scale ranging from 0 (not at all) to 4 (extremely). Higher scores represent higher intensity of distress during the past week.

SECONDARY OUTCOMES:
Change in Perceived stress | Baseline, 8 weeks (post-intervention for experimental group), 16 weeks (follow-up for experimental group, post-intervention for control group)
  Perceived stress will be assessed with the Perceived Stress Scale-4 (Warting et al., 2013). The questions in this scale ask you about your feelings and thoughts related to stress during the last month, with 0 representing "seldom" and 4 representing "very often." Higher scores are correlated to more stress.
Change in Posttraumatic stress | Baseline, 8 weeks (post-intervention for experimental group), 16 weeks (follow-up for experimental group, post-intervention for control group)
  The PTSD CheckList - Civilian Version (PCL-C) will be used to assess PTSD symptoms (Ruggiero et al., 2003). The PCL is a self-report scale for PTSD comprising 17 items that correspond to the key symptoms of PTSD. Respondents indicate how much they have been bothered by a symptom over the past month using a 5-point (1-5) scale, with high scores characterize higher intensity of PTSD.
Change in Adherence to Medication Assisted Treatment (MAT) | Baseline, 8 weeks (post-intervention for experimental group), 16 weeks (follow-up for experimental group, post-intervention for control group)
  Adherence to other medical treatments not given as part of this study will be assessed with the Adherence to Refills and Medications Scale (ARMS; Kripalani et al., 2009). The ARMS scale is a 12 item scale that measures adherence to medications.
Change in Mindfulness skills | Baseline, 8 weeks (post-intervention for experimental group), 16 weeks (follow-up for experimental group, post-intervention for control group)
  FFMQ-15: 15-item Five-Facet Mindfulness Questionnaire https://www.sussexpartnership.nhs.uk/sites/default/files/documents/jenny_gus_short_ffmq-15_june_16.pdf. The FFMQ-15 measures 5 subscales of mindfulness: Observing, Describing, Acting with Awareness, Non-judgement, Non-reactivity; Scores range from 15 to 75, with higher scores indicating higher levels of mindfulness skills.
Change in Perceived Quality of Life (health, well-being) | Baseline, 8 weeks (post-intervention for experimental group), 16 weeks (follow-up for experimental group, post-intervention for control group)
  Quality of life will be assessed with the World Health Organization Quality of Life (WHOQOL-BREF; World Health Organization, 2004). The 26-item scale assesses quality of life, health, and other areas of wellbeing. Items are measured on a five-point scale. Higher scores represent higher quality of life.
Change in Extent of mindfulness self-practice | Baseline, 8 weeks (post-intervention for experimental group), 16 weeks (follow-up for experimental group, post-intervention for control group)
  Participants will be asked the following questions: "Besides the sessions you may have attended as part of this study, on your own, 'Did you engage in mindfulness meditation or other mindfulness practices in the past two months (8 weeks)?', 'How many days per week did you engage in mindfulness meditation or other mindfulness practices?', 'How long in minutes did you meditate per session of mindfulness meditation?', 'Describe your practice of mindfulness (what exercises/activities/techniques did you practice?).'" For quantitative analyses, we will use the variable representing number of days of mindfulness practice per week. We will also assess the number of sessions attended, number of non-completers, and reasons for dropout.
Change in Frequency of major depressive disorder relapse episodes | Baseline, 8 weeks (post-intervention for experimental group), 16 weeks (follow-up for experimental group, post-intervention for control group)
  The number of Major depressive relapse episodes will be identified using the ICD-10 codes for MDD in the DSM-5 (First, 2014).

OTHER OUTCOMES:
Change in Emotion regulation | Baseline, 8 weeks (post-intervention for experimental group), 16 weeks (follow-up for experimental group, post-intervention for control group)
  Emotion regulation will be assessed with the Difficulties in Emotion Regulation Scale-Short Form (Kaufman et al., 2016), an 18-item measure used to identify emotional regulation issues in adults. Higher values reflect greater difficulty with emotion regulation
Change in Savoring | Baseline, 8 weeks (post-intervention for experimental group), 16 weeks (follow-up for experimental group, post-intervention for control group)
  The Savoring Beliefs Inventory (Bryant, 2003) is a 24-item questionnaire consisting of three subscales: anticipating, savoring the moment, and reminiscing. Half of the items are positively formulated, while the other half are negatively framed. Each item is rated on a 7-point Likert scale ranging from "strongly disagree" to "strongly agree." Higher scores indicate higher levels of savoring.
Intervention fidelity | Intervention fidelity will be assessed over the course of 8 weeks for each intervention group cohort.
  Intervention fidelity will be assessed with the Mindfulness-Based Relapse Prevention Adherence and Competence Scale (MBRP-AC; Chawla et al., 2010). All sessions will be audio recorded. Two members of the research team will rate 50% of a random selection of sessions using the MBRP-AC. Raters will code at least 10 practice sessions, which will be reviewed with the research team until acceptable reliability is achieved, and they will attend regular recalibration meetings to prevent drift. Group facilitators will also meet weekly with the licensed clinical psychologist, a member of the research team, for supervision.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Shi, Ph.D., Principal Investigator — Clemson University
Locations (2):
- United States (2):
  - Clemson University, Clemson, South Carolina
  - Prisma Health, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared outside the research team.

REFERENCES:
- [Background] Ames CS, Richardson J, Payne S, Smith P, Leigh E. Mindfulness-based cognitive therapy for depression in adolescents. Child Adolesc Ment Health. 2014 Feb;19(1):74-78. doi: 10.1111/camh.12034. Epub 2013 Aug 28. PMID 32878358
- [Background] Baer RA, Smith GT, Lykins E, Button D, Krietemeyer J, Sauer S, Walsh E, Duggan D, Williams JM. Construct validity of the five facet mindfulness questionnaire in meditating and nonmeditating samples. Assessment. 2008 Sep;15(3):329-42. doi: 10.1177/1073191107313003. Epub 2008 Feb 29. PMID 18310597
- [Background] Batink T, Peeters F, Geschwind N, van Os J, Wichers M. How does MBCT for depression work? studying cognitive and affective mediation pathways. PLoS One. 2013 Aug 23;8(8):e72778. doi: 10.1371/journal.pone.0072778. eCollection 2013. PMID 24009704
- [Background] Bryan F. Savoring Beliefs Inventory (SBI): A scale for measuring beliefs about savouring. Journal of Mental Health. 2003; 12(2):175-196.
- [Background] Căzănescu, DG, Tecuta, L, Cândea, DM, & Szentagotai-Tătar, A. Savoring as mediator between irrational beliefs, depression, and joy. Journal of Rational-Emotive & Cognitive-Behavior Therapy. 2019; 37(1): 84-95.
- [Background] Chawla N, Collin S, Bowen S, Hsu S, Grow J, Douglass A, Marlatt GA. The mindfulness-based relapse prevention adherence and competence scale: development, interrater reliability, and validity. Psychother Res. 2010 Jul;20(4):388-97. doi: 10.1080/10503300903544257. PMID 20204916
- [Background] Derogatis LR, Melisaratos N. The Brief Symptom Inventory: an introductory report. Psychol Med. 1983 Aug;13(3):595-605. PMID 6622612
- [Background] Hanson HM, Salmoni AW. Stakeholders' perceptions of programme sustainability: findings from a community-based fall prevention programme. Public Health. 2011 Aug;125(8):525-32. doi: 10.1016/j.puhe.2011.03.003. Epub 2011 Jul 29. PMID 21802700
- [Background] Kaufman EA, Xia M, Fosco G, Yaptangco M, Skidmore CR, Crowell, SE. The Difficulties in Emotion Regulation Scale Short Form (DERS-SF): Validation and replication in adolescent and adult samples. Journal of Psychopathology and Behavioral Assessment. 2016; 38(3), 443-455.
- [Background] IsHak WW, Greenberg JM, Balayan K, Kapitanski N, Jeffrey J, Fathy H, Fakhry H, Rapaport MH. Quality of life: the ultimate outcome measure of interventions in major depressive disorder. Harv Rev Psychiatry. 2011 Sep-Oct;19(5):229-39. doi: 10.3109/10673229.2011.614099. PMID 21916825
- [Background] Joormann J, Stanton CH. Examining emotion regulation in depression: A review and future directions. Behav Res Ther. 2016 Nov;86:35-49. doi: 10.1016/j.brat.2016.07.007. Epub 2016 Jul 28. PMID 27492851
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Merikangas KR, Walters EE. Lifetime prevalence and age-of-onset distributions of DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):593-602. doi: 10.1001/archpsyc.62.6.593. PMID 15939837
- [Background] Kessing LV, Hansen MG, Andersen PK, Angst J. The predictive effect of episodes on the risk of recurrence in depressive and bipolar disorders - a life-long perspective. Acta Psychiatr Scand. 2004 May;109(5):339-44. doi: 10.1046/j.1600-0447.2003.00266.x. PMID 15049770
- [Background] Kripalani S, Risser J, Gatti ME, Jacobson TA. Development and evaluation of the Adherence to Refills and Medications Scale (ARMS) among low-literacy patients with chronic disease. Value Health. 2009 Jan-Feb;12(1):118-23. doi: 10.1111/j.1524-4733.2008.00400.x. PMID 19911444
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Kuyken W, Watkins E, Holden E, White K, Taylor RS, Byford S, Evans A, Radford S, Teasdale JD, Dalgleish T. How does mindfulness-based cognitive therapy work? Behav Res Ther. 2010 Nov;48(11):1105-12. doi: 10.1016/j.brat.2010.08.003. Epub 2010 Aug 13. PMID 20810101
- [Background] Lengacher CA, Kip KE, Reich RR, Craig BM, Mogos M, Ramesar S, Paterson CL, Farias JR, Pracht E. A Cost-Effective Mindfulness Stress Reduction Program: A Randomized Control Trial for Breast Cancer Survivors. Nurs Econ. 2015 Jul-Aug;33(4):210-8, 232. PMID 26477119
- [Background] Lorant V, Croux C, Weich S, Deliege D, Mackenbach J, Ansseau M. Depression and socio-economic risk factors: 7-year longitudinal population study. Br J Psychiatry. 2007 Apr;190:293-8. doi: 10.1192/bjp.bp.105.020040. PMID 17401034
- [Background] Ma SH, Teasdale JD. Mindfulness-based cognitive therapy for depression: replication and exploration of differential relapse prevention effects. J Consult Clin Psychol. 2004 Feb;72(1):31-40. doi: 10.1037/0022-006X.72.1.31. PMID 14756612
- [Background] MacKenzie MB, Kocovski NL. Mindfulness-based cognitive therapy for depression: trends and developments. Psychol Res Behav Manag. 2016 May 19;9:125-32. doi: 10.2147/PRBM.S63949. eCollection 2016. PMID 27274325
- [Background] Mason O, Hargreaves I. A qualitative study of mindfulness-based cognitive therapy for depression. Br J Med Psychol. 2001 Jun;74(Pt 2):197-212. PMID 11453171
- [Background] Mathers CD, Loncar D. Projections of global mortality and burden of disease from 2002 to 2030. PLoS Med. 2006 Nov;3(11):e442. doi: 10.1371/journal.pmed.0030442. PMID 17132052
- [Background] Michalak J, Holz A, Teismann T. Rumination as a predictor of relapse in mindfulness-based cognitive therapy for depression. Psychol Psychother. 2011 Jun;84(2):230-6. doi: 10.1348/147608310X520166. Epub 2011 Apr 13. PMID 22903859
- [Background] Mueller TI, Leon AC, Keller MB, Solomon DA, Endicott J, Coryell W, Warshaw M, Maser JD. Recurrence after recovery from major depressive disorder during 15 years of observational follow-up. Am J Psychiatry. 1999 Jul;156(7):1000-6. doi: 10.1176/ajp.156.7.1000. PMID 10401442
- [Background] Piet J, Hougaard E. The effect of mindfulness-based cognitive therapy for prevention of relapse in recurrent major depressive disorder: a systematic review and meta-analysis. Clin Psychol Rev. 2011 Aug;31(6):1032-40. doi: 10.1016/j.cpr.2011.05.002. Epub 2011 May 15. PMID 21802618
- [Background] Ruggiero KJ, Del Ben K, Scotti JR, Rabalais AE. Psychometric properties of the PTSD Checklist-Civilian Version. J Trauma Stress. 2003 Oct;16(5):495-502. doi: 10.1023/A:1025714729117. PMID 14584634
- [Background] Segal ZV, Williams M, & Teasdale J. (2018). Mindfulness-based cognitive therapy for depression. Guilford Publications.
- [Background] Sharplin GR, Jones SB, Hancock B, Knott VE, Bowden JA, Whitford HS. Mindfulness-based cognitive therapy: an efficacious community-based group intervention for depression and anxiety in a sample of cancer patients. Med J Aust. 2010 Sep 6;193(S5):S79-82. doi: 10.5694/j.1326-5377.2010.tb03934.x. PMID 21542452
- [Background] Stirman SW, Miller CJ, Toder K, Calloway A. Development of a framework and coding system for modifications and adaptations of evidence-based interventions. Implement Sci. 2013 Jun 10;8:65. doi: 10.1186/1748-5908-8-65. PMID 23758995
- [Background] Warttig SL, Forshaw MJ, South J, White AK. New, normative, English-sample data for the Short Form Perceived Stress Scale (PSS-4). J Health Psychol. 2013 Dec;18(12):1617-28. doi: 10.1177/1359105313508346. Epub 2013 Oct 22. PMID 24155195
- [Background] World Health Organization. (2008). The global burden of disease: 2004 update. World Health Organization.
- [Background] World Health Organization. (2004). The world health organization quality of life (WHOQOL)- BREF (No. WHO/HIS/HSI Rev. 2012.02). World Health Organization.
- [Background] First, M. B. (2014). "Structured Clinical Interview for the DSM (SCID)." In The Encyclopedia of Clinical Psychology, edited by Robin L. Cautin and Scott O. Lilienfeld, 26:1-6. Hoboken, NJ, USA: John Wiley & Sons, Inc.
- [Background] Gross, J. J., & Thompson, R. A. (2006). Emotion regulation: Conceptual foundations. Handbook of emotion regulation.
- [Derived] Hooshmand Zaferanieh M, Shi L, Jindal M, Chen L, Zhang L, Lopes S, Jones K, Wang Y, Meggett K, Walker CB, Falgoust G, Zinzow H. Web-Based Mindfulness-Based Cognitive Therapy for Adults With a History of Depression: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Jun 18;13:e53966. doi: 10.2196/53966. PMID 38888958